CLINICAL TRIAL: NCT00685711
Title: An Escalating Single Intradermal or Subcutaneous Dose Study in Cat Allergic Subjects to Assess the Safety of Cat-PAD.
Brief Title: Safety of Cat-PAD in Cat Allergic Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Responsible Party: Rod Hafner, Circassia Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP001
Record Dates: First submitted 2008-05-20; First posted 2008-05-28 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Cat Allergy
Keywords: Cat allergy; Immunotherapy; Cat-PAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Placebo intradermal n = 2 with each dose level of Cat-PAD.
  Interventions: Biological: Cat-PAD
- 2 (Experimental): Intradermal injection of increasing single doses of Cat-PAD (0.03, 0.3, 3, 12 nmol) n = 6 per dose level. Based on review of blinded LPSR, an additional dose of Cat-PAD between 0.03 and 12 nmol may be administered to an additional cohort of 6 subjects.
  Interventions: Biological: Cat-PAD
- 3 (Placebo Comparator): Placebo subcutaneous n = 2 with each dose level of Cat-PAD.
  Interventions: Biological: Cat-PAD
- 4 (Experimental): Subcutaneous injection of increasing single doses of Cat-PAD (0.03, 0.3, 3, 12, 20 nmol) n = 6 per dose level. Based on review of blinded LPSR, an additional dose of Cat-PAD between 0.03 and 20 nmol may be administered to an additional cohort of 6 subjects.
  Interventions: Biological: Cat-PAD

INTERVENTIONS:
Biological: Cat-PAD — single, escalating dose intradermal and subcutaneous injections of Cat-PAD

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma. Cat-PAD is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of cat allergy. This study will investigate the safety of Cat-PAD administered as increasing single doses.

DETAILED DESCRIPTION:
This study is designed as a two centre, randomised, placebo-controlled, escalating single dose study in up to 88 cat allergic subjects. Cohorts of 8 subjects will be enrolled. Each cohort will undergo screening 14-28 days before treatment and a baseline challenge for EPSR and LPSR to cat allergen injected into the arm 7 days before treatment. On the treatment day, subjects will be injected either intradermally (into the skin) or subcutaneously (under the skin) with a single dose of Cat-PAD or placebo and safety observations made for 8 h. After 21 days, subjects will again have cat allergen injected into the arm and the EPSR and LPSR will be recorded. The dose of Cat-PAD will be increased in successive cohorts, provided that the previous dose tested was well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* A reliable history of rhinoconjunctivitis (sneezing, rhinorrhoea, nasal blockage, itchy/red/sore/watering eyes) or controlled asthma (GINA (2006) classification 1) on exposure to cats for at least 1 year.
* Late-Phase Allergic Skin Reaction (LPSR) to 0.010 HEP units Leti cat allergen eight hours after intradermal injection of greater than 25mm diameter response on single arm.

Exclusion Criteria:

* Subjects with asthma falling under GINA(2006) classification 2 (partly controlled) and 3 (uncontrolled).
* A history of anaphylaxis to cat allergen.
* Subjects with a cat specific IgE >100 kU/L.
* Subjects with an FEV1 <80% of normal.
* Subjects with an acute phase skin response to cat allergen with a weal diameter > 30mm.
* Subjects who suffer from hay fever, and cannot complete the clinical study outside the pollen season.
* Allergen immunotherapy during the last 5 years or Cat Dander immunotherapy ever.
* Use of the following therapies for the periods specified prior to the screening visit will make the subject ineligible for the study: corticosteroids: (depot: 90 days; systemic: 30 days; dermatological, intranasal, inhalational: 15 days); cromones (14 days); antihistamines other than loratadine (nasal and long-acting oral: 10 days; short-acting oral, ocular: 7 days); leukotriene inhibitors (10 days); anticholinergics (7 days); alpha-adrenergic agonists (7 days); tricyclic antidepressants (14 days). If it becomes a medical necessity for a subject to use one of these contraindicated medications during the study this will become an individual stopping criteria.
* Subjects for whom administration of adrenaline is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* Subjects being treated with beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Cat-PAD | 0, 7, 21 days

SECONDARY OUTCOMES:
Late-Phase Skin Reaction (LPSR) 8 hours after intradermal challenge with whole cat allergen. | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, MD Professor, Principal Investigator — Allergy-Centre-Charité
Locations (1):
- Allergy-Centre-Charité, Berlin, Germany